CLINICAL TRIAL: NCT02218996
Title: Treatment of Anxiety Disorders for Children and Adolescents in Regular Outpatient Clinics (TADCAROC)
Brief Title: Treatment of Anxiety Disorders for Children and Adolescents in Regular Outpatient Clinics
Acronym: TADCAROC
Status: Active, not recruiting | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Helse Vest (Other)
Responsible Party: Sponsor
Other Study IDs: ID416
Record Dates: First submitted 2014-08-08; First posted 2014-08-18 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Anxiety Disorders
Keywords: Anxiety; Children; Adolescent; Effectiveness; Outpatient
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Psychosocial treatment: Children and adolescents with anxiety disorders
  Interventions: Other: Psychosocial treatment

INTERVENTIONS:
Other: Psychosocial treatment — Regular psychosocial treatment in clinical outpatient service.

SUMMARY:
The purpose of this study is to examine the content of the treatment being delivered for anxiety disorders for children and adolescents in the regular outpatient clinics in western Norway. The study will also collect data before and after treatment to evaluate the result of the treatment. Furthermore, as part of the study we aim to collect normative data on two questionnaires used to identify anxiety symptoms and the extent to which anxiety interfere with daily functioning. We also aim to develop a quality indicator for anxiety treatment that can be used to monitor treatment in the regular outpatient service, based on the results of the current study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of an anxiety disorder (including PTSD and OCD) based on the diagnostic interview ADIS (ADIS-C/P; Silverman & Albano, 1996).
* The anxiety disorder is the patients primary diagnosis.
* Informed concent is given.

Exclusion Criteria:

* The patient is in need for other primary treatment intervention (e.g., psychosis, suicidality risk)

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children/adolescents from 7-17 years old referred to ordinary outpatient mental health service.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The Anxiety Disorder Interview Schedule for Diagnostic and Statistical Manual (DSM-IV), child and parent versions (ADIS- C/P; Silverman & Albano, 1996). | The primary outcome measure will be administered pre-treatment, post treatment (an expected average of 20 weeks) and at ten year follow-up.
  Diagnostic interview for anxiety disorders and other comorbid disorders. For the 10-year follow-up we anticipate to use another version of the diagnostic interview schedule based on revised diagnostic criteria for anxiety disorders.

SECONDARY OUTCOMES:
Children's Anxiety Life Interference Scale (CALIS; Lyneham et al., 2013) | This outcome measure will be administered pre-treatment and post treatment (an expected average of 20 weeks).
The Screen for Child Anxiety Related Emotional Disorders (SCARED; Birmaher et al., 1999). | This outcome measure will be administered pre-treatment and post treatment (an expected average of 20 weeks).
Spence Children's Anxiety Scale (SCAS; Spence, 1998) | This outcome measure will be administered pre-treatment and post treatment (an expected average of 20 weeks).
The Strengths and Difficulties Questionnaire (SDQ; Goodman, 1997) | This outcome measure will be administered pre-treatment and post treatment (an expected average of 20 weeks)
Short Mood & Feeling Questionaire (SMFQ; Angold et al., 1995). | This outcome measure will be administered pre-treatment and post treatment (an expected average of 20 weeks)
Clinical Global Impressions (CGI; Guy, 1976). | The outcome measure will be administered pre-treatment, post treatment (an expected average of 20 weeks) and at ten year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jon F Bjaastad, D. Psych, Principal Investigator — Division of Psychiatry, Stavanger University Hospital, N-4068 Stavanger, Norway
Locations (1):
- BUPA Helse Stavanger, Stavanger, Rogaland, Norway

IPD SHARING:
Plan to Share IPD: No